CLINICAL TRIAL: NCT01611389
Title: Minimizing Right Ventricular Pacing in Dual-chamber Pacemaker Patients With Sinus Node Disease and First Degree Atrioventricular Block.
Brief Title: Minimizing Ventricular Pacing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Military Institute od Medicine National Research Institute (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 83562; N N402 533539 (Other Grant/Funding Number: National Science Centre)
Record Dates: First submitted 2012-05-31; First posted 2012-06-05 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-05

CONDITIONS: Sinus Node Disease.; First Degree Atrioventricular Block.
MeSH Terms: conditions — Sick Sinus Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Long AV delay. (Experimental)
  Interventions: Device: Prolonging atrioventricular (AV) delay.
- Short AV delay. (Active Comparator)
  Interventions: Device: Standard atrioventricular (AV) delay.

INTERVENTIONS:
Device: Prolonging atrioventricular (AV) delay. — Prolonging atrioventricular (AV) delay to maximum 350 ms.
  Arms: Long AV delay.
Device: Standard atrioventricular (AV) delay. — Standard atrioventricular (AV) delay - approximately 180/140 ms depending on heart rate.
  Arms: Short AV delay.

SUMMARY:
The aim of this study is to evaluate the effect of minimizing right ventricular pacing in dual-chamber pacemaker patients with sinus node disease (SND) and first degree atrioventricular block (AVIB)on exercise capacity, quality of life and other heart failure measures.

ELIGIBILITY:
Inclusion Criteria:

* prolonged PQ interval > 200 ms,
* percentage of right ventricular pacing with standard AV delay > 90.

Exclusion Criteria:

* second or third degree atrioventricular block,
* permanent atrial fibrillation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Oxygen uptake (cardiopulmonary exercise testing). | 3 months

SECONDARY OUTCOMES:
Left ventricular ejection fraction. | 3 months
  Assessed in echocardiography.
Quality of life | 3 months
  SF36 questionnaire.
Arrhythmia | 3 months
  24 hours Holter monitoring, pacemaker storage data.
Ventilatory anaerobic threshold (cardiopulmonary exercise testing) | 3 months
VE/VCO2 slope (cardiopulmonary exercise testing). | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Military Institute of Medicine, Warsaw, Poland